CLINICAL TRIAL: NCT03720951
Title: Comparison Between Applying Pulsed Radiofrequency to the Pudendal Nerve Bilaterally Vs Its Application to Sacral Nerve Roots S2,3 and 4 Bilaterally in the Improvement of Pain and Symptoms in Chronic Prostatitis, A Prospective Randomized Study
Brief Title: Applying Pulsed Radiofrequency to the Pudendal Nerve Bilaterally Vs Its Application to Sacral Nerve Roots S2,3 and 4 Bilaterally in Chronic Prostatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Radio frequency prostatitis
Record Dates: First submitted 2018-10-20; First posted 2018-10-26 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Prostatitis; Pulsed Radiofrequency
Keywords: Pulsed Radiofrequency; chronic Prostatitis
MeSH Terms: conditions — Prostatitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I(Pudendal n.) (Experimental): Fluoroscopic-guided pulsed R.F. to pudendal nerve bilaterally under image guidance
  Interventions: Radiation: pudendal nerve
- Group II(Sacral n.) (Experimental): Fluoroscopic-guided pulsed R.F. to nerve roots S 2, 3, 4 bilaterally under image guidance
  Interventions: Radiation: sacral n roots

INTERVENTIONS:
Radiation: pudendal nerve — Fluoroscopic-guided pulsed R.F. to pudendal nerve bilaterally under image guidance
  Arms: Group I(Pudendal n.)
Radiation: sacral n roots — Fluoroscopic-guided pulsed R.F. to nerve roots S 2, 3, 4 bilaterally under image guidance
  Arms: Group II(Sacral n.)

SUMMARY:
Prevalence estimates show that prostatitis is one of the most common urological conditions and that symptoms range considerably among men of various socioeconomic status, race, and age. For men under 50 years, prostatitis is the most common urologic outpatient diagnosis. Chronic prostatitis/chronic pelvic pain syndrome has high prevalence estimates internationally ( 16% North America, 14% Asian & Europeans). Men suffering from Chronic prostatitis/chronic pelvic pain syndrome report significant impairment in their quality of life which is also associated with greater health care expenditures.

DETAILED DESCRIPTION:
The hallmark indicator of Chronic prostatitis/chronic pelvic pain syndrome has been identified as enduring pain in the perineum, pelvic area, and/or genitalia in many studies. As in other painful chronic conditions, pain does not correspond strongly with objective medical findings and has no orthodox pathology. It is however associated with voiding and sexual disturbances. Symptoms should have been present for at least 3 months within the previous 6 months and must be validated with the standard questionnaire of the National Institute of Health-Chronic Prostatitis Symptom Index. In most patients, pain is the main symptom. Chronic bacterial prostatitis the predominant type of prostatitis is a common and painful condition, typified by pelvic area pain and lower urinary tract symptoms, for which effective diagnostic techniques and treatment strategies remain elusive. Previous studies have documented an association between prostatitis and both psychiatric and rheumatologic diseases. Socioeconomic status indicators, such as lower education and lower income, also played an important role in predicting which men would have worse chronic prostatitis symptoms. These findings are consistent with those found among women with interstitial cystitis; women with lower education and income in the Interstitial Cystitis Database were more likely to report more severe symptoms.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III.

Exclusion Criteria:

* those with infection at the site of injection,
* coagulopathy or another bleeding diathesis,
* a pre-existing neurologic deficit in the targeted region,

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score | after 1 month of the intervention
  Visual Analogue Score for pain rating( 0 = no pain(minimum) and 10 = the most severe pain(maximum)) will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

REFERENCES:
- [Background] Cahana A, Van Zundert J, Macrea L, van Kleef M, Sluijter M. Pulsed radiofrequency: current clinical and biological literature available. Pain Med. 2006 Sep-Oct;7(5):411-23. doi: 10.1111/j.1526-4637.2006.00148.x. PMID 17014600
- [Background] Issa W, Roumeguere Te, Bossche MV. [Chronic pelvic pain syndrome]. Rev Med Brux. 2013 Jan-Feb;34(1):29-37. French. PMID 23534312
- [Background] Pontari M, Giusto L. New developments in the diagnosis and treatment of chronic prostatitis/chronic pelvic pain syndrome. Curr Opin Urol. 2013 Nov;23(6):565-9. doi: 10.1097/MOU.0b013e3283656a55. PMID 24080807